CLINICAL TRIAL: NCT03424616
Title: Deep Brain Stimulation of Nucleus Accumbens for Opioid Relapse Prevention:A Multicenter Randomized Double-Blind Sham-stimulation Controlled Clinical Trial
Brief Title: Deep Brain Stimulation of Nucleus Accumbens for Opioid Relapse Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: National Institute on Drug Dependence, Peking University (Unknown); Ruijin Hospital (Other); West China Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAcDBSORP
Record Dates: First submitted 2018-01-17; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Addiction
Keywords: Opiate dependence; Deep brain stimulation; Nucleus accumbens
MeSH Terms: conditions — Behavior, Addictive; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Stagger-on design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative immediate Deep brain stimulation (Experimental): The addicts undergone the deep brain stimulation while the stimulation (Suzhou Sceneray® DBS System) was turned on 1-2 weeks postoperatively.
  Interventions: Device: Suzhou Sceneray® DBS System
- Postoperative delayed Deep brain stimulation (Sham Comparator): The addicts undergone the deep brain stimulation while the stimulation (Suzhou Sceneray® DBS System) was off until 25 months postoperatively, during which the following up was kept, then the the stimulation was turned on 25 months postoperatively.
  Interventions: Device: Suzhou Sceneray® DBS System

INTERVENTIONS:
Device: Suzhou Sceneray® DBS System — We plan to use the SceneRay 1242 (SceneRay, SuZhou, China) electrode with a diameter of 1.27 mm and 4 contacts. The SceneRay 1242 electrode combined with the SceneRay 1181 implantable pulse generator has the advantage of adaptive coverage area for the Ventral Capsule/Ventral Striatum, enabling simultaneous implantation in the nucleus accumbens (NAc; 2 ventral contacts) and the anterior limb of the internal capsule (ALIC; 2 dorsal contacts) with independently programmed parameters such as frequency, amplitude, and voltage; and remote and wireless programing, which allows for convenient and prompt adjustments in emergency situations.

SUMMARY:
Nucleus accumbens plays important roles in the process of opiate addiction and initial of relapse after detoxification.According to the single-centered preliminary open-labeled prospective trial results, the investigators hypothesize that bilateral stimulation of the NAc will effectively reduce the relapse of the opiate dependence.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old < Age < 50 years old
* Moderate to severe opiates abuse disorders (fulfilled diagnostic-criteria according to DSM-5)

  1. History of opiates abuse no less than 3 years
  2. Failure of at least three addiction treatments ( in hospital or compulsive rehabilitation）, among which failure of methadone maintenance treatment must be met
  3. completion of detoxification ( Negative urine test for morphine, methamphetamine, ketamine and buprenorphine)
* Free patient's decision/informed Consent (existing comprehensive ability in meaning, methodology and execution of the study and ability of acceptance, known the benefit and risk of the treatment)

Exclusion Criteria:

* Clinical relevant psychiatric comorbidity (schizophrenic psychoses, bipolar affective diseases, severe personality disorder)
* Contraindications of a MRI-examination, e.g. implanted cardiac pacemaker/heart defibrillator
* Abuse of other type of drugs
* severe cognitive impairments
* Enrollment in other clinical trials
* Stereotactic respectively neurosurgical intervention in the past
* Contraindications of a stereotactic operation, e.g. increased bleeding-disposition, cerebrovascular diseases (e.g. arteriovenous malfunction, aneurysms, systemic vascular diseases)
* Serious and instable organic diseases (e.g. instable coronal heart disease)
* tested positively for HIV
* pregnancy and/or lactation
* Severe disorders for coagulation and liver function
* Epilepsy or other severe brain trauma or neurological impairments

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-06 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
The abstinent rate at 25 weeks after DBS stimulation on （Urine Tests） | At 25 weeks after DBS stimulation on
  If the participants or their families report no less than 2 times of the drug use in each of two consecutive weeks, or the consecutive 2 times of urine tests showed positive, or lost of follow-up, the case was defined as relapse

SECONDARY OUTCOMES:
The total days of abstinence for participants | Baseline (preoperative), 4 weeks, 12 weeks, 25 week after DBS stimulation on
  The total days of abstinence for participants
The longest duration for sustained abstinence for participants | Baseline (preoperative), 4 weeks, 12 weeks, 25 week after DBS stimulation on
  The longest duration for sustained abstinence for participants
Visual analog scale (VAS) craving score for opioid drugs | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  Ranging from 0-10,with 0 indicates no craving while 10 indicates extreme craving
Body weight for participants | Baseline (preoperative), 4 weeks, 12 weeks, 25 week after DBS stimulation on
  Body weight for participants
Hamilton Depression Scale（HAMD-17) | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  17 items,Total scores<7: normal;7<Total scores<17:possible depression;17<Total scores<24:definite depression;Total score>24: severe depression
Scaling for Opiate withdrawal symptoms | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  There were 19 items for rating 19 withdrawl symptoms, with 0 indicating none and 4 indicating most severe, the total scores are obtained by summary for scores of each items, ranging from 0-76, the higher the total scores indicating the worsen opiate withdrawl symptoms.
The evaluation on MATRICS-test | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  Software system constructed by MATRICS company, which was used for evaluate the cognitive function of the participants
The rate of positive urine test results | Baseline (preoperative), 4 weeks, 12 weeks, 25 week after DBS stimulation on
  times of positive urine test/ total times of urine test
Hamilton Anxiety Scale (HAMA) | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  14 items, Total scores<6: normal;7<Total scores<14:possible anxiety;14<Total scores<21:definite anxiety;Total score>21: severe anxiety
Pittsburgh sleep quality index(PSQI) | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  Scaling for evaluating the sleep quality, the higher total scores indicating the more difficulties on sleep, thus the higher total scores indicating the worsen sleep quality
Fagerstrom Test Nicotine Dependence assessment (FTND) | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  Scaling for Nicotine Dependence: The higher of scores indicating higher lever of Nicotine Dependence
Social Disability Screening Schedule (SDSS) | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  Scaling for Social Disability with 10 items, the higher total scores indicating the much severe social disability
Activity of Daily Living Scale (ADL) | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  Consists of Physical Self-maintenance Scale and Instrumental Activities of Daily Living Scale, ranging from 0-56, total scores <14, normal; total score >14, ADL dysfunction
36-Item Short Form Health Survey (SF-36) | Baseline (preoperative), 1week, 4 weeks, 12 weeks, 25 week after DBS stimulation on
  Scaling for Quality of life with 8 subscales, the higher total scores indicating the better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Guodong Gao, M.D., Principal Investigator — Department of neurosurgery, Tangdu Hospital; Lin Lu, M.D., Principal Investigator — National Institute on Drug Dependence, Peking University
Locations (5):
- China (5):
  - National Institute on Drug Dependence, Peking University, Beijing, Beijing Municipality
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Department of neurosurgery, Tangdu Hospital, Xi'an, Shaanxi
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan

REFERENCES:
- [Derived] Qu L, Ge S, Li N, Wang W, Yang K, Wu P, Wang X, Shi J. Clinical evaluation of deep brain stimulation of nucleus accumbens/anterior limb of internal capsule for opioid relapse prevention: protocol of a multicentre, prospective and double-blinded study. BMJ Open. 2019 Feb 13;9(2):e023516. doi: 10.1136/bmjopen-2018-023516. PMID 30765398